CLINICAL TRIAL: NCT00551811
Title: A Dose Ranging Study to Assess the Effect of Pre-treatment With a Single Dose of Oral SB656933 on Lung Inflammation Following Challenge With Inhaled Ozone and Intermittent Exercise in Healthy Volunteers, Relative to Placebo
Brief Title: Evaluate the Effects of the Drug (SB-656933-AAA) on the Body After a Single Dose in Subjects Who Have Inhaled Ozone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: CR2100597
Record Dates: First submitted 2007-10-29; First posted 2007-10-31 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: SB-656933-AAA,; ozone challenge; single dose,
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Subjects receiving treatment sequence 1 (Experimental): Eligible subjects will receive single doses of placebo in period 1, SB-656933-AAA with a dose of 50 milligrams in period 2 and 150 milligrams in period 3.
  Interventions: Drug: SB-656933-AAA; Drug: Placebo
- Subjects receiving treatment sequence 2 (Experimental): Eligible subjects will receive single doses of SB-656933-AAA with a dose of 50 milligrams in period 1, placebo in period 2 and SB-656933-AAA 150 milligrams in period 3.
  Interventions: Drug: SB-656933-AAA; Drug: Placebo
- Subjects receiving treatment sequence 3 (Experimental): Eligible subjects will receive single doses of SB-656933-AAA with a dose of 50 milligrams in period 1, 150 milligrams in period 2 and placebo in period 3.
  Interventions: Drug: SB-656933-AAA; Drug: Placebo

INTERVENTIONS:
Drug: SB-656933-AAA — SB-656933-AAA tablets will be available with a dose strength of 50 milligrams, administered orally.
Drug: Placebo — Placebo tablets will be intended to be administered orally.

SUMMARY:
A study to evaluate the effect of SB-656933-AAA on the body after a single dose in subjects who have been challenged with ozone.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects between 18-50 years.
* Females should be of non-child bearing potential.
* Non-smoking for at least 12 months.
* Normal lung function.
* Subjects should be able to produce acceptable sputum samples.

Exclusion Criteria:

* Any serious medical condition.
* Hepatitis B or C and/or HIV positive.
* Currently on regular medication except paracetamol.
* Body Mass Index <20 or >30.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2007-10-08 (Actual); Primary Completion 2008-07-22 (Actual); Study Completion 2008-07-22 (Actual)

PRIMARY OUTCOMES:
To assess the effect of a single dose of SB-656933-AAA on ozone-induced inflammation in healthy subjects. Total number of neutrophils in sputum 6 hours after inhaling ozone. | 6 hours after inhaling ozone

SECONDARY OUTCOMES:
Total number of white cells in sputum 6 hours after inhaling ozone. Concentration of protein in sputum. Safety of SB-656933-AAA. | 6 hours after inhaling ozone

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Berlin, Germany

REFERENCES:
- [Background] Lazaar AL, Sweeney LE, MacDonald AJ, Alexis NE, Chen C, Tal-Singer R. SB-656933, a novel CXCR2 selective antagonist, inhibits ex vivo neutrophil activation and ozone-induced airway inflammation in humans. Br J Clin Pharmacol. 2011 Aug;72(2):282-93. doi: 10.1111/j.1365-2125.2011.03968.x. PMID 21426372
- See also: Results for study CR2100597 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/CR2100597?search=study&study_ids=CR2100597#rs